CLINICAL TRIAL: NCT00664625
Title: Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of BMS-791325 in Subjects Chronically Infected With Hepatitis C Virus Genotype 1
Brief Title: A Single Ascending Dose Study of BMS-791325 in HCV Infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI443-002
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): BMS-791325 (100 mg)
  or
  placebo match for (100 mg)
  Interventions: Drug: BMS-791325; Drug: Placebo
- 2 (Experimental): BMS-791325 (300 mg)
  or
  placebo match for (300 mg)
  Interventions: Drug: BMS-791325; Drug: Placebo
- 3 (Experimental): BMS-791325 (900 mg)
  or
  placebo match for (900 mg)
  Interventions: Drug: BMS-791325; Drug: Placebo
- 4 (Experimental): BMS-791325 (potential dose between 10-800 mg)
  or
  placebo match for (10-800 mg)
  Interventions: Drug: BMS-791325; Drug: Placebo

INTERVENTIONS:
Drug: BMS-791325 — Capsules, Oral, Once Daily, Single Dose
Drug: Placebo — Capsules, Oral, Once Daily, Single Dose

SUMMARY:
The primary purpose of this study is to evaluate the safety profile and tolerability of single oral doses of BMS-791325 in subjects with chronic hepatitis C infection

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected with HCV genotype 1
* Treatment naive or treatment non-responders or treatment intolerant
* HCV RNA viral load of ≥10*5* IU/mL
* BMI 18 to 35 kg/m²

Exclusion Criteria:

* Any significant acute or chronic medical illness which is not stable or is not controlled with medication and not consistent with HCV infection
* Major surgery within 4 weeks of study drug administration and any gastrointestinal surgery that could impact the absorption of study drug
* Co-infection with HIV or HBV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measures | Safety and tolerability assessments will be performed for a period of 7 days after administration of a single dose

SECONDARY OUTCOMES:
Pharmacokinetic Measures | Pharmacokinetic assessments will be done for a period of 72 hours following administration of a single oral dose
Pharmacodynamic Measures | Antiviral activity will be assessed by the magnitude and rate of change in plasma HCV RNA levels for a period of 7 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (5):
  - Advanced Clinical Res Inst, Anaheim, California
  - West Coast Clinical Trials, Llc, Cypress, California
  - Washington University School Of Medicine, St Louis, Missouri
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Alamo Medical Research, San Antonio, Texas
- Local Institution, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Sims KD, Lemm J, Eley T, Liu M, Berglind A, Sherman D, Lawitz E, Vutikullird AB, Tebas P, Gao M, Pasquinelli C, Grasela DM. Randomized, placebo-controlled, single-ascending-dose study of BMS-791325, a hepatitis C virus (HCV) NS5B polymerase inhibitor, in HCV genotype 1 infection. Antimicrob Agents Chemother. 2014 Jun;58(6):3496-503. doi: 10.1128/AAC.02579-13. Epub 2014 Apr 14. PMID 24733462
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx